CLINICAL TRIAL: NCT04630392
Title: Effects of the Addition of a Single Bout of Whole-Body Vibration to a Single Bout of Treadmill Training on Gait and Spasticity in Ambulatory Children With Cerebral Palsy
Brief Title: Effects of Treadmill Training and Whole-body Vibration in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Jianhua Wu, Associate Professor, Georgia State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H19180
Record Dates: First submitted 2020-09-25; First posted 2020-11-16 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Self-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): There are two intervention groups: treadmill walking only, whole-body vibration plus treadmill walking.
  Interventions: Other: Treadmill Training; Other: Whole Body Vibration & Treadmill Training

INTERVENTIONS:
Other: Treadmill Training — Ten minutes of treadmill walking at 110% self-selected overground walking speed
Other: Whole Body Vibration & Treadmill Training — Eight bouts of 90 seconds of vibration at 20 Hz and an amplitude of 2 mm on a Galileo Med-L side-to-side-alternating WBV plate (StimDesigns LLC, Carmel, CA, USA) followed by ten minutes of treadmill walking at 110% self selected overground walking speed.

SUMMARY:
Whole-body vibration (WBV) and treadmill training (TT) are commonly-utilized rehabilitation interventions for children with neuromotor disorders. WBV has been shown in the literature to positively affect gait and lower body spasticity in this population. However, the effects of a single session of WBV are generally transient, lasting between ten minutes and two hours. Thus, it may be necessary to combine WBV with another intervention to reinforce improved movement patterns and maximize its potential benefits. Therefore, the aim of this study is to investigate the effects of the addition of a single bout of WBV to a single bout of TT on the lower extremity spasticity and gait parameters of ambulatory children with CP.

DETAILED DESCRIPTION:
Whole-body vibration (WBV) and treadmill training (TT) are commonly-utilized rehabilitation interventions for children with neuromotor disorders. The evidence supporting the use of TT in children with cerebral palsy (CP) remains inconclusive, but WBV has been shown in the literature to positively affect gait and lower body spasticity in this population. However, the effects of a single session of WBV are generally transient, lasting between ten minutes and two hours. Thus, it may be necessary to combine WBV with another intervention to reinforce improved movement patterns and maximize its potential benefits. Therefore, the aim of this study is to investigate the effects of the addition of a single bout of WBV to a single bout of TT on the lower extremity spasticity and gait parameters of ambulatory children with CP.

The investigators plan to recruit 20 children between the ages of 6 and 17 with spastic CP. Subjects will complete a 10-minute bout of TT at 110% of their preferred overground (OG) walking speed, rest for 15 minutes, and then complete a 12-minute bout of WBV at 20Hz and 2mm followed by a second 10-minute bout of TT at the same speed. OG gait characteristics, including spatiotemporal parameters, joint kinematics, and electromyographic (EMG) parameters, will be collected at 5 time points: before the first bout of TT, immediately following the first bout of TT, before WBV, immediately following WBV, and immediately following the second bout of TT. Lower extremity spasticity will be assessed using multiple methods at the same time points. Changes in gait parameters and spasticity will be assessed using a one-way repeated measures ANOVA and a series of dependent t-tests. Significant level will be set at α = 0.05.

The investigators anticipate that acute improvements in OG gait parameters will be greater following the combined bout of WBV and TT than the bout of TT alone. The investigators expect this to be due to the reduction of lower extremity spasticity following WBV, which should allow for more normalized gait patterns during TT and improve carryover to OG gait. Further, the investigators expect to gain insight into the mechanisms responsible for spasticity reduction following WBV which will allow for the making of informed decisions regarding clinical rehabilitative protocols involving WBV and TT.

ELIGIBILITY:
Inclusion Criteria:

* a medical diagnosis of spastic CP
* a GMFCS level of I, II, or III
* age of 6-17 years at the time of data collection

Exclusion Criteria:

* history of musculoskeletal injury within the past 3 months
* history of Botox injections to the lower extremities within the past 3 months
* history of significant cardiac abnormalities and/or uncontrolled seizures
* any cognitive or behavioral issues that prevent the subject from safely following instructions while walking on the treadmill

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overground gait walking speed | immediately after intervention
  Measured in m/s from kinematic motion capture data
Overground gait step length | immediately after intervention
  Measured in cm from kinematic motion capture data
Overground gait dynamic knee range of motion | immediately after intervention
  Measured in degrees from kinematic motion capture data
Overground gait dynamic ankle range of motion | immediately after intervention
  Measured in degrees from kinematic motion capture data
Overground gait muscle activity as measured by electromyographic sensors | immediately after intervention
  integrated area per gait cycle at the following muscles: biceps femoris, vastus lateralis, lateral gastrocnemius, tibialis anterior
Lower extremity spasticity as measured by the Modified Tardieu Test | immediately after intervention
  including R1 and R2 joint angles as well as qualitative score

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Wu, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No